CLINICAL TRIAL: NCT02736097
Title: A Multicenter Study to Evaluate Predictive Factors for Multidrug Resistant Healthcare Associated Pneumonia in Critically Ill Patients
Brief Title: Drug Resistance Factors In Healthcare-associated Pneumonia
Acronym: DEFINE
Status: Completed | Type: Observational
Sponsor: Critical Care Pharmacotherapy Trials Network (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Ishaq Lat, Primary Investigator, Critical Care Pharmacotherapy Trials Network
Other Study IDs: 15071001
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Pneumonia; Critical Illness
MeSH Terms: conditions — Pneumonia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently clinical guidelines categorize pneumonia in to three types: community, healthcare-associated, and hospital-acquired. Much of the existing research to describe the epidemiology of pneumonia in critically ill patients comes from single-center studies or from retrospective database analyses, which limit generalizability and lead to over-prescription of broad-spectrum antibacterial agents. This will be a prospective, multicenter epidemiological study to characterize pneumonia epidemiology in critically ill adult patients.

DETAILED DESCRIPTION:
Pneumonia is one of the leading causes of death in the United States and is associated with significant costs to the healthcare system. Recent treatment guidelines describe a new subtype of pneumonia, healthcare-associated pneumonia (HCAP), to identify those patients who present to a hospital from the community and are thought to be at greater risk for developing pneumonia due to multidrug resistant organisms (MDRO).

The HCAP categorization scheme is intended to improve the prescription of initial appropriate empiric antibacterial agents and minimize the morbidity and mortality associated with inappropriate empiric selection.However, one of the chief criticisms of the guideline recommendations is that the criteria used to define HCAP is overly broad, which may result in greater use of broad-spectrum antibiotics.

The prevailing notion is that many patients in the community will be at the lowest risk for experiencing MDR pneumonia and can be treated with a less broad anti-infective regimen. Patients with increasing exposure to the healthcare system will receive initial anti-infective therapy that is more broad in an effort to target MDROs. The investigator group believes that it is not simply exposure to the healthcare system that predicts the incidence of MDR pneumonia (i.e., criteria for HCAP), but rather, the "intensity" of exposure to the healthcare system that is predictive of MDR pneumonia. The aim of this study is to identify risk factors for MDR HCAP pneumonia in critically ill patients. .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* ICU admission
* Empiric or directed anti-infective treatment for pneumonia for ≥ 5 days

Exclusion Criteria:

* Patient stay in ICU for < 24 hours
* Patient transfer to the ICU from a hospital floor following prescription for anti-infective therapy in the previous 24 hours of ICU admission
* Diagnosis of cystic fibrosis or bronchiectasis
* Fungal pneumonia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to an intensive care unit requiring anti-infective therapy for the traetment of pneumonia.
Sampling Method: Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of multidrug resistant pneumonia pathogen | 30 days

SECONDARY OUTCOMES:
Incidence of pneumonia subtypes | 30 days

CONTACTS AND LOCATIONS:
Locations (30):
- United States (29):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Hartford Healthcare, Hartford, Connecticut
  - University of Florida - Jacksonville Hospital, Jacksonville, Florida
  - Cleveland Clinic - Florida, Weston, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Roudebush - Indianapolis Veterans Administration Hospital, Indianapolis, Indiana
  - University of Kentucky Healthcare - Chandler Medical Center, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - University of Minnesota - Fairview Health Services, Minneapolis, Minnesota
  - Northeast Regional Medical Center, Kirksville, Missouri
  - Lakes Regional General Healthcare, Laconia, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Mercy Medical Center, Canton, Ohio
  - Cleveland Clinic - Cleveland, Cleveland, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Healthcare Family, Austin, Texas
  - Memorial Hermann Healthcare System, Houston, Texas
  - University of Wisconsin Hospital, Madison, Wisconsin
  - Medical College of Wisconsin/ Froedtert Hospital, Milwaukee, Wisconsin
- Ministry of of National Guard-Health Affaires, Riyahd, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lat I, Daley MJ, Shewale A, Pangrazzi MH, Hammond D, Olsen KM; DEFINE study group and the Discovery Research Network. A Multicenter, Prospective, Observational Study to Determine Predictive Factors for Multidrug-Resistant Pneumonia in Critically Ill Adults: The DEFINE Study. Pharmacotherapy. 2019 Mar;39(3):253-260. doi: 10.1002/phar.2171. Epub 2018 Oct 3. PMID 30101412